CLINICAL TRIAL: NCT05637827
Title: The Initiating Factors of Myopia Among Primary and Secondary School Students in Tianjin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tianjin children myopia
Record Dates: First submitted 2022-11-26; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children with hyperopia: The refractive error and axial length of eye were observed
  Interventions: Other: No intervention
- children with emmetropia: The refractive error and axial length of eye were observed
  Interventions: Other: No intervention
- children with myopia: The refractive error and axial length of eye were observed
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention in each group, and only the natural development was observed

SUMMARY:
There was a prospective cohort observational study. Forty hyperopic children, 40 myopic children and 120 emmetropia children were randomly selected from grade 1 to grade 3, and were followed up every six months for 3 years. All patients received cycloplegic refraction examination, ocular biological test, binocular visual function test and a questionnaire related to daily eye habits. A multi-level and multi-dimensional data analysis model was constructed to explore the possible factors affecting the occurrence and development of myopia in children.

ELIGIBILITY:
Inclusion Criteria:

* students in grades 1-3
* Can cooperate with the examination of students

Exclusion Criteria:

* Obvious strabismus and amblyopia
* Eye diseases that affect vision, such as congenital cataracts, glaucoma, and retinal diseases
* History of ocular surgery

Ages: 5 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Healthy children with hyperopia, emmetropia and myopia
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of refractive error | Every 6 months for a period 3 years
  The changes of refractive error between visit time in every 6 months
The changes of axial length | Every 6 months for a period 3 years
  The changes of axial length between visit time in every 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Result] Rose KA, French AN, Morgan IG. Environmental Factors and Myopia: Paradoxes and Prospects for Prevention. Asia Pac J Ophthalmol (Phila). 2016 Nov/Dec;5(6):403-410. doi: 10.1097/APO.0000000000000233. PMID 27898443
- [Result] Seidemann A, Schaeffel F. An evaluation of the lag of accommodation using photorefraction. Vision Res. 2003 Feb;43(4):419-30. doi: 10.1016/s0042-6989(02)00571-0. PMID 12535999